CLINICAL TRIAL: NCT00473486
Title: A Randomized (PhaseII), Double-blind, Multicenter Phase I/II Trial of Pemetrexed, Carboplatin Plus or Minus Sorafenib in the First-line Treatment of Patients With Stage IIIb or IV Non-Small Cell Lung Cancer
Brief Title: Study in Patients With Advanced Non-Small Cell Lung Cancer Treated With Pemetrexed and Carboplatin Plus or Minus Sorafenib
Acronym: PECASO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sorafenib administered in the combination with pemetrexed-carboplatin appears to enhance thrombocytopenia compared to historical data.
Sponsor: University Hospital Muenster (Other)
Collaborators: Bayer (Industry); Eli Lilly and Company (Industry)
Responsible Party: Dr. Christian Brandts Principal Investigator, University Hospital Muenster and University Hospital of Frankfurt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-005970-26; KKS / INNERE_A / NSCLC2006
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2007-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pemetrexed, Carboplatin plus Sorafenib in the first-line treatment of patients with stage IIIb or IV NSCLC
  Interventions: Drug: pemetrexed, carboplatin, sorafenib
- 2 (Placebo Comparator): Pemetrexed, Carboplatin plus placebo in the first-line treatment of patients with stage IIIb or IV NSCLC
  Interventions: Drug: pemetrexed, carboplatin, placebo

INTERVENTIONS:
Drug: pemetrexed, carboplatin, sorafenib — Ph. 1: pemetrexed 500mg/m² iv day 1; carboplatin AUC 6 iv day 1; Sorafenib 200mg po bid days 2-19; 400mg po bid days 2-19
  Ph 2: pemetrexed 500mg/m² iv day 1; carboplatin AUC 6 iv day 1;sorafenib depending on results of Ph 1
  Arms: 1
Drug: pemetrexed, carboplatin, placebo — Ph 2: pemetrexed 500mg/m² iv day 1; carboplatin AUC 6 iv day 1; placebo day 2-19
  Arms: 2

SUMMARY:
The majority of patients with advanced NSCLC treated with standard platinum based chemotherapy regimens ultimately develop disease progression. Active therapies with improved toxicity profiles are clearly needed in this setting. The primary objective of this trial is to assess the toxicity profile and to determine the effect on progression free survival and time to progression in patients with advanced NSCLC treated with sorafenib in addition to carboplatin and pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Locally advanced (stage IIIB with malignant pleural or pericardial effusion) or metastatic (stage IV) NSCLC
* No prior systemic chemotherapy
* Prior local radiotherapy is allowed if it is completed at least 3 weeks prior to the first dose of study medication; also concomitant palliative radiotherapy to an existing bone lesion for pain control is allowed
* Prior surgery is allowed if it is performed at least 4 weeks prior to the first dose of study medication and patient should be fully recovered.
* Must have measurable disease with at least one lesion with a longest diameter measured as ≥ 2 cm with conventional techniques or as ≥ 1 cm with spiral CT
* Age ≥18 years old
* ECOG performance score (PS) 0-1
* Life expectancy of at least 12 weeks
* Adequate bone marrow, renal and hepatic function

  * hemoglobin ≥ 9.0 g/dl
  * absolute neutrophil count ≥1,500/mm3
  * platelet count ≥ 100,000/mm3
  * total bilirubin ≤ 1.5 times the upper limit of normal
  * ALT and AST ≤ 2.5 times the upper limit of normal (≤ 5 x upper limit of normal for patients with liver involvement)
  * INR ≤ 1.5 and aPTT within normal limits
  * serum creatinine ≤ 1.5 the upper limit of normal
* Patients with creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing patients
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least six months after the last administration of sorafenib
* Signed informed consent prior to any study specific procedures
* Compliance and geographic proximity that allow adequate follow-up

Exclusion Criteria:

* Any prior systemic anticancer therapy including cytotoxic therapy, targeted agents, experimental therapy (treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study enrollment), adjuvant, or neo-adjuvant therapy for NSCLC
* Any participation in a clinical trial 30 days prior to study entry and concomitantly to the study
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (angina symptoms at rest) or new-onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
* Documented brain metastases (unless the patient is > 6 months from definitive therapy for brain metastases, has a negative imaging study within 4 weeks of study entry and has been off corticosteroids for at least 4 weeks before study enrolment). Brain imaging (CT scan/MRI) is required in symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients.
* Patients with seizure disorder requiring medication (such as steroids or antiepileptics)
* Known HIV infection or chronic hepatitis B or C
* Active clinically serious infections > CTCAE Grade 2
* Presence of clinically significant third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study enrolment
* Pulmonary hemorrhage/bleeding event >= CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event > =Grade 3 within 4 weeks of first dose of study drug
* Evidence or history of bleeding diathesis or coagulopathy
* Therapeutic anticoagulation with vitamin K antagonists such as phenprocoumon, warfarin, or with heparins or heparinoids. Low dose anticoagulation is permitted
* Serious, non-healing wound, ulcer, or bone fracture
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug
* Known or suspected allergy to sorafenib, carboplatin or pemetrexed
* Previous or current cancer that is distinct in primary site or histology from NSCLC except cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis) or any cancer curatively treated > 3 years prior to study entry
* Substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study
* Significant weight loss (> or equal 10% body weight during preceeding 6 weeks)
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose ≤ 1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam)
* Inability or unwillingness to take folic acid, vitamin B12 supplementation or corticosteroids
* Recent (within 30 days of enrolment) or concurrent yellow fever vaccination
* Serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Ph.1: Identify the recommended phase II dose of sorafenib for combination therapy with carboplatin and pemetrexed | July 2008
Ph.2: Compare the PFS of carboplatin/pemetrexed + sorafenib or carboplatin/pemetrexed + placebo in patients with stage IIIb or IV non-small cell lung cancer | May 2009

SECONDARY OUTCOMES:
Ph.1: Determine dose limiting toxicity | July 2008
Ph 1: Determine the safety profile of the combination treatment | July 2008
Ph 1: descriptive analysis of efficacy | July 2008
Ph.2: Compare PFS of carboplatin/pemetrexed + sorafenib or carboplatin/pemetrexed + placebo in patients with stage IIIb or IV NSCLC | May 2009
Ph 2: Assess time to progression in patients treated with either regimen | May 2009
Ph 2: Determine the overall survival in patients treated with either regimen | May 2009
Ph 2: Determine the objective response rate (CR, PR), disease control rate (CR,PR,SD), time to response and duration of response | May 2009
Ph 2: Identify surrogate markers from the tumor biopsy or resection specimen from the time of diagnosis that predict response | May 2009
Ph 2: Assess Quality of Life of patients treated with either regimen | May 2009
Ph 2: Assess feasibility and toxicity profile of this regimen | May 2009

CONTACTS AND LOCATIONS:
Overall Officials: Christian Brandts, MD, Principal Investigator — Universitätsklinikum Münster, Med. Klinik und Poliklinik A, Hämatologie, Onkologie und Pneumologie and Uniklinik Frankfurt Innere Medizin, Hämatologie/Onkologie, 60590 Frankfurt
Locations (1):
- University of Muenster, Dept. of Medicine, Hematology / Oncology, Münster, Germany